CLINICAL TRIAL: NCT02097784
Title: Interest of the Echocardiography in the Management of Cirrhotic Patients With Acute Kidney Injury
Acronym: CIRREN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013.831; 2013-A01622-43 (Other: ANSM)
Record Dates: First submitted 2014-03-24; First posted 2014-03-27 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Cirrhosis; Hepatorenal Syndrome; Acute Kidney Injury; Diastolic Function
Keywords: cirrhosis; hepatorenal syndrome; acute kidney injury; diastolic function
MeSH Terms: conditions — Fibrosis; Hepatorenal Syndrome; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cirrhosis with portal hypertension,ascite and acute kidney (Other)
  Interventions: Procedure: Echocardiography

INTERVENTIONS:
Procedure: Echocardiography

SUMMARY:
This prospective study focuses on the interest of the echocardiography for cirrhotic patients, who present acute kidney injury corresponding to the criteria of hepatorenal syndrome. This echocardiography will be done before the volemic expansion and the final diagnostic of hepatorenal syndrome or prerenal azotemia. The primary endpoint is to describe the hemodynamic characteristics of this population at the time of acute kidney injury and their association with diagnostic of hepatorenal syndrome or prerenal azotemia. Patients with elevated filling pressure, predicting poor outcome of volemic expansion will be excluded of the study after the echocardiography and will not undergo volemic expansion but appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* patients > 18 years
* written consent for the participation of the study
* cirrhosis with portal hypertension and ascite
* acute kidney injury according to AKIN criteria (rapid increase of creatinine (48 hours) > 26.4 µmol or > 50% comparing with baseline). Baseline creatinine is the last value of creatinine before admission or creatinine at the admission if stable during 5 days.
* absence of argument for acute tubular necrosis or other organic acute renal injury
* absence of argument for shock

Exclusion Criteria:

* pregnant women
* volemic expansion before echocardiography
* portal thrombosis
* presence of TIPSS
* history of cardiac or renal pathology
* atrial fibrillation
* cardiac valvulopathy
* technical limitation due to echogenicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Hemodynamic features assessed by echocardiography before the volemic expansion of cirrhotic patients with acute renal injury corresponding to the criteria of hepatorenal syndrome. | At Day0 : at the time of diagnostic of acute kidney injury, before volemic expansion.
  Systolic and diastolic function assessment, filling pressures, pulmonary arterial hypertension

SECONDARY OUTCOMES:
Tolerance of volemic expansion, as recommended by international guidelines | After 48 hours of volemic expansion
  Clinical tolerance of volemic expansion, acute pulmonary oedema
Response to vasoconstrictor treatment of hepatorenal syndrome, in case of diagnostic of hepatorenal syndrome | 1 month after inclusion
  Renal function recovery, renal replacement therapy, liver transplantation
Mortality | 1 month after inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Fanny LEBOSSE, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon, France